CLINICAL TRIAL: NCT02525328
Title: Genome Study in Constitutional Thinness
Acronym: GENOSCANN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0908129; 2010-A00051-38 (Other: ANSM)
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Thinness; Leanness
Keywords: Constitutional Thinness; linkage study; genome wide scan (GWAS)
MeSH Terms: conditions — Thinness | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood or saliva specimen in families including at least one well phenotyped CT index case (grade 2 or 3 of thinness according WHO classification). Family's members are : CT subjects and subjects without CT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CT subjects: blood or saliva specimen
  Interventions: Other: blood or saliva specimen
- subjects without CT: blood or saliva specimen
  Interventions: Other: blood or saliva specimen

INTERVENTIONS:
Other: blood or saliva specimen — blood or saliva specimen is sampled for DNA extraction in CT family's members

SUMMARY:
Constitutional thinness (CT) is a recently defined entity as a differential diagnosis of anorexia nervosa (AN), considered to be the most frequent cause of low body mass index (BMI) in young women. CT subjects present no AN psychiatric traits, preserved menses, no biological signs of undernutrition and balanced energy metabolism despite a Body Mass Index (BMI) <17 kg / m².

CT familial aggregation, low body mass without a hormonal explanation, and specific appetite regulation profile suggest a specific genetic profile in these subjects.

Objective: A family linkage study in order to identify genes involved in the constitutional thinness phenotype by using genome wide scan (GWAS) techniques Studied population: Fifty families including at least one well phenotyped CT index case (grade 2 or 3 of thinness according WHO classification). Blood or saliva is sampled for DNA extraction.

Perspectives: Revealing eventual abnormalities could lead to a more precise diagnosis of constitutional thinness and new hypothesis in understanding extreme bodyweight mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* For all subjects:

  * age > 18 yrs
  * affiliation to health insurance
  * member of a family including at least 2 CT members and overall 3 evaluable members over 2 generations
  * written and signed consent
* For CT subjects :

  * grade 2 or 3 of thinness according WHO classification
  * women, BMI < 17 kg/m² at 20-30 yrs or < 19 for older subjects
  * men, BMI < 18 kg/m² at 20-30 yrs or < 20 for older subjects
  * absence of DSM criteria for anorexia nervosa
  * young women : normal menses and fat mass percentage 15 % ; absence of DSM criteria for anorexia nervosa
  * men : normal testosterone level
* For subjects without CT :

  * women, BMI > 19 kg/m²
  * men, BMI > 20 kg/m²

Exclusion Criteria:

* CT subjects:

  * smoking > 5 cigarettes / day
  * history of emaciating pathologies
  * intense physical activity > 7 hours / week
* For all subjects :

  * refuse of written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifty families including at least 2 well phenotyped CT index case (grade 2 or 3 of thinness according WHO classification) and members without CT.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2010-10-21 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
chromosome regions' abnormalities | day 1
  The linkage study is performed in order to identify one or several chromosome regions linked the constitutional thinness phenotype by using genome wide scan (GWAS) techniques in CT families members.

SECONDARY OUTCOMES:
genetic markers | day 1
  Identify within upper mentioned regions more specific genetic markers (mutation/variant) to characterize genes involved in CT phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Estour, MD PhD, Principal Investigator — CHU SAINT-ETIENNE; Bogdan GALUSCA, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No